CLINICAL TRIAL: NCT02433613
Title: Postmarket Evaluation of the Phased Radio Frequency Ablation System (GOLD AF Registry)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Collaborators: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: GOLD AF
Record Dates: First submitted 2015-03-17; First posted 2015-05-05 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: Pulmonary Vein Isolation; Phased Radiofrequency Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, multi-center, single-arm, non-interventional and open-label registry. The purpose of the registry is to document use of Phased Radio Frequency Ablation (RFA) (hereafter "Phased RFA") System in a real world patient population with atrial fibrillation (AF) and evaluate its performance.

Gold AF will enroll a minimum of 1,000 patients who undergo Phased RFA in approximately 38 sites in Western, Central Europe, Israel and South Korea.

DETAILED DESCRIPTION:
This registry will collect data prospectively on patients with paroxysmal, persistent and longstanding persistent atrial fibrillation (hereafter "AF") undergoing Phased RFA treatment. Phased RFA will be applied according to the 'Intended Use' in CE mark (European Conformity) release and product packaging.

The treatment will be performed according to routine hospital practice and no additional tests are required specific to the registry. This registry will serve as a tool to collect clinical data in order to expand the knowledge base of safety, effectiveness and functionality of the Medtronic Phased RFA System in a real world patient population.

The key measures collected for the patients will be inclusive of, but are not limited to, clinical data pertaining to AF and individual disease state(s) characterized by form of AF and underline diseases, Phased RFA procedure details including timing and catheters in use, procedure and system related adverse events, AF recurrence, re-ablations and left atrial flutter rate after the index Phased RFA procedure. Additionally, this study will provide further information in the evolving anticoagulation strategies (e.g. continuous versus bridging and vitamin K antagonist versus novel oral anticoagulants) in the setting of AF ablations. Patients will be followed minimum for 12 months and maximum for 14 months after the Phased RFA ablation procedure. The twelve month follow-up can be done by telephone if it is not standard of care in the hospital's practice. During the twelve month follow-up patients will be interviewed with a quality of life questionnaire and results will be compared to the quality of life questionaire completed before the procedure.

ELIGIBILITY:
Inclusion criteria:

* Patient with AF who is scheduled for Phased RFA procedure
* Patient signed patient informed consent or patient data release form
* Age ≥18 years old To avoid enrollment bias in this cohort of patient and reflect "real world" clinical practice for Phased RFA no exclusion criteria will be defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible are all patients with paroxysmal, persistent and long-standing persistent AF who fulfill all inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1071 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Boersma, MD, Ph.D, Principal Investigator — St. Antonious; Meleze Hocini, MD, Principal Investigator — Hôpital Cardiologique du Haut-Lévêque
Locations (41):
- France (4):
  - CHU Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CMC Parly 2, Le Chesnay
  - Centre Cardiologique du Nord, Saint-Denis
- Jo Ann Medical Center, Tbilisi, Georgia
- Germany (6):
  - St. Johannes Hospital, Dortmund
  - Evangelisches Krankenhaus, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Herz- und Gefäßzentrum Oberallgäu-Kempten, Kempten
  - Universitätsklinikum Münster, Münster
  - St. Vincenz-Krankenhaus Paderborn, Paderborn
- General Hospital Alexandra, Athens, Greece
- Hungary (2):
  - Military Hospital, Budapest
  - University of Debrecen, Debrecen
- Israel (4):
  - The Barzilai Medical Center Ashkleon, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Hadassah Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
- Italy (5):
  - A.O. Papa Giovanni XXIII, Bergamo
  - Az. Osped. Pugliese Ciaccio, Catanzaro
  - Ospedale Mater Salutis, Legnago
  - A.O. Osped. S.Gerardo, Monza
  - A.O. San Camillo Forlanini, Rome
- Netherlands (2):
  - Medisch Centrum Leeuwarden B.V., Leeuwarden
  - St. Antonius Ziekenhuis, Nieuwegein
- Poland (4):
  - Samodzielny Publiczny Szpital Kliniczny Nr 4, Lublin
  - Samodzielny Publiczny Szpital Kliniczny Nr 2, Szczecin
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
  - 4 Wojskowy Szpital Kliniczny, Wroclaw
- Centro Hospitalar Lisboa Notre - Hospital de Santa Maria E.P.E., Lisbon, Portugal
- South Korea (6):
  - Sejong General Hospital, Bucheon-si
  - Keimyung University Dongsan Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Hirslanden Klinik St. Anna AG, Zurich, Switzerland
- Eastbourne District General Hospital, Eastbourne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Phased RFA System: Observation study / registry with one patient group. Data on the use of the Phased AF system in the "real world" clinical practice / daily routine of EP (electrophysiology) laboratories utilizing the Phased AF system was collected.
Period: Overall Study
Arm/Group | Phased RFA System
Started | 1071
Completed | 1054
Not Completed | 17

BASELINE CHARACTERISTICS:
Groups:
- Phased RFA System: Observation study / registry with one patient group. Data on the use of the Phased AF system in the "real world" clinical practice / daily routine of EP laboratories utilizing the Phased AF system was collected.
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1054
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341
  Male | 713
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hungary | 37
  United Kingdom | 6
  Portugal | 57
  Switzerland | 33
  Spain | 73
  Greece | 9
  Netherlands | 181
  South Korea | 73
  Poland | 123
  Italy | 182
  Israel | 40
  Georgia | 2
  France | 42
  Germany | 213
Body-Mass-Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.8 (4.5)
Atrial Fibrillation (AF) Status [Count of Participants; unit: Participants]
  Paroxysmal Atrial Fibrillation (PAF) | 740
  Persistent Atrial Fibrillation | 279
  Longstanding persistent Atrial Fibrillation | 35
Symptomatic Atrial Fibrillation [Count of Participants; unit: Participants] | 1007

OUTCOME MEASURES:

1. Primary Outcome: Estimate Phased RFA (Radio Frequency Ablation) Mid-term Success Rate
Description: Success rate will be estimated as time to first event: AF recurrence and/or left Atrial Flutter. Parameters of interest include: re-ablations, ECG/EGM (electrogram) recorded AF, electrical and pharmacological cardioversions.
Time Frame: Patient will be followed for minimum 12 months, maximum 14 months after index Phased RFA
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1054
Days | 185.1 (76.6)

2. Secondary Outcome: Estimate Phased RFA Mid-term Safety
Description: Estimate major procedure/system related complications of Phased RFA
Time Frame: Patient will be followed for minimum 12 months, maximum 14 months after index Phased RFA
Measure: Number; unit: events
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1054
events | 27

3. Other Pre Specified Outcome: Acute Procedural Success Rate
Description: Procedure considered successful if all PVs (pulmonary veins) were isolated (entrance and/or exit block confirmation per vein) and procedure was not declined due to technical issues related to Phased RFA system
Time Frame: Patient will be followed in the Catheterization Laboratory (hereafter "CathLab")/operating room during approximately 2 hours of Phased RFA procedure duration
Measure: Number; unit: % of procedural success rate
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1036
% of procedural success rate | 94.3

4. Other Pre Specified Outcome: Procedural Efficiency - Procedure Duration, Laboratory Occupancy Duration and Fluoroscopy Time
Description: Parameters to measure the efficiency: procedure duration, laboratory occupancy duration, fluoroscopy time
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1048
Minutes
  General Procedure Time | 107.0 (39.5)
  Duration of PVAC ablation | 58.0 (28.8)
  Time from delivery to cathlab to 3D Mapping | 171.1 (66.1)
  Cathlab Occupancy Time | 154.7 (49.3)
  Total Fluoroscopy Time | 25.0 (15.5)

5. Other Pre Specified Outcome: Peri-procedural Anticoagulation Therapy - Activated Clotting Time
Description: Characterize anticoagulation therapy: activated clotting time (ACT) during the procedure. Correlate anticoagulation therapy with thromboembolic events and bleeding the peri -procedural thromboembolic events and bleeding
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1054
seconds
  Highest activated clotting time (ACT) | 356.9 (115.7)
  Lowest ACT | 274.4 (95.3)

6. Other Pre Specified Outcome: Single Catheter PVAC (Pulmonary Vein Ablation Catheter) GOLD Utilization in Persistent AF Ablation - Phased RFA Catheters Used
Description: Evaluate which tools participating centers use (MAAC (Multi-Array Ablation Catheter) and/or MASC (Multi-Array Septal Catheter) and/or PVAC GOLD) in persistent and long standing persistent AF and to verify patient's characteristics, procedure approaches and estimates outcome across participating sites. The main interest is if PVAC GOLD catheter can be utilized as a single catheter for patients with persistent AF and analyze AF recurrence rate in this group
Time Frame: Patient will be followed for minimum 12 months, maximum 14 months after index Phased RFA
Population: Patients with persistent AF only
Measure: Mean (Standard Deviation); unit: catheter
Arm/Group | Phased RFA System
Number analyzed (Participants) | 279
catheter | 2.1 (1.1)

7. Other Pre Specified Outcome: Quality of Life Dynamic - AFEQT Score at 12 Months
Description: Quality of life will be captured using the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire. It is a standardized, disease-specific, reliable and responsive measure of health-related quality of life in subjects with AF. The AFEQT is a self-reported questionnaire with responses on a 7-point Likert scale. The 20-item instrument is divided into three domains (4-item symptom score, 8-item daily activities score, 6-item treatment concerns score) plus two treatment satisfaction questions.In countries where no validated version is available yet (e.g. Israel, Portugal), the AFEQT questionnaire will not be applied or will be additionally validated for the country official languages according to local requirements and regulations.
  Overall or subscale range from 0 to 100. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability).
Time Frame: Patient will be followed for minimum 12 months, maximum 14 months, 12 month reported
Population: 911 patients filled in validated language versions of the AFEQT; 143 patients filled in not validated language versions; AFEQT score at baseline available for 954 patients. The response on the AFEQT are scored on a 1 to 7 Likert scale, 1 = "not at all" to 7 = "Extremely".
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1054
score on a scale
  AFEQT Score at Baseline: number analyzed (Participants) | 954
  AFEQT Score at Baseline | 56.6 (20.3)
  AFEQT Score at 12 Months Follow-Up (site visit): number analyzed (Participants) | 204
  AFEQT Score at 12 Months Follow-Up (site visit) | 82.6 (18.0)
  AFEQT Score at 12 Months Follow-Up (phone call): number analyzed (Participants) | 499
  AFEQT Score at 12 Months Follow-Up (phone call) | 85.4 (18.6)
  Changes in QoL Score Baseline to 12 M FU (visit): number analyzed (Participants) | 199
  Changes in QoL Score Baseline to 12 M FU (visit) | 24.5 (23.0)
  Changes in QoL Score Baseline to 12 M FU (phone): number analyzed (Participants) | 459
  Changes in QoL Score Baseline to 12 M FU (phone) | 29.1 (24.9)

8. Other Pre Specified Outcome: Procedural Efficiency - Number of Catheters Used
Description: Parameters to measure the efficiency: Phased RFA consumables used
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: catheters
Units Other Than Participants: procedures
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1048
Number analyzed (procedures) | 1054
catheters | 2.2 (1.3)

9. Other Pre Specified Outcome: Procedural Efficiency - Number of Adjunctive Devices Used
Description: Parameters to measure the efficiency: adjunctive devices used
Time Frame: as for outcome 3
Measure: Number; unit: procedures
Units Other Than Participants: procedures
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1048
Number analyzed (procedures) | 1054
procedures | 209

10. Other Pre Specified Outcome: Peri-procedural Anticoagulation Therapy - International Normalized Ratio (INR)
Description: Characterize anticoagulation therapy: international normalized ratio (INR). Correlate anticoagulation therapy with thromboembolic events and bleeding the peri -procedural thromboembolic events and bleeding. The INR is derived from prothrombin time (PT) which is calculated as a ratio of the patient's PT to a control PT standardized for the potency of the thromboplastin reagent developed by the World Health Organization (WHO) using the following formula: INR = Patient PT ÷ Control PT. INR can be used to assess the risk of bleeding or the coagulation status of the patients.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1054
ratio | 1.4 (0.6)

11. Other Pre Specified Outcome: Peri-procedural Anticoagulation Therapy - Percent of Participants With Previous and Peri-Procedural Anticoagulation Therapy
Description: Characterize anticoagulation therapy: utilization of vitamin K antagonists (VKA), novel oral anticoagulants (NOAC), peri -procedural "bridging" vs "no bridging" strategy. Correlate anticoagulation therapy with thromboembolic events and bleeding the peri -procedural thromboembolic events and bleeding
Time Frame: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Phased RFA System
Number analyzed (Participants) | 1054
percentage of patients
  Oral anticoagulants discontinued before procedure | 53.8
  Previously treated with VKA | 23.2
  Previously treated with NOACs | 63.5
  Major procedure related event (stroke) | 0.2

12. Other Pre Specified Outcome: Single Catheter PVAC (Pulmonary Vein Ablation Catheter) GOLD Utilization in Persistent AF Ablation - Number Total Cardioversions
Description: as for outcome 6
Time Frame: Patient will be followed for minimum 12 months, maximum 14 months after index Phased RFA
Population: Patients with persistent AF only
Measure: Mean (Standard Deviation); unit: cardioversions
Arm/Group | Phased RFA System
Number analyzed (Participants) | 279
cardioversions | 3.0 (1.0)

13. Other Pre Specified Outcome: Single Catheter PVAC (Pulmonary Vein Ablation Catheter) GOLD Utilization in Persistent AF Ablation - Percentage of Persistent AF Participants With Cardioversions for AF Within Last 12 Months
Description: as for outcome 6
Time Frame: as for outcome 3
Population: Patients with persistent AF only
Measure: Number; unit: percentage of persistent AF patients
Arm/Group | Phased RFA System
Number analyzed (Participants) | 279
percentage of persistent AF patients | 71.0

14. Other Pre Specified Outcome: Single Catheter PVAC (Pulmonary Vein Ablation Catheter) GOLD Utilization in Persistent AF Ablation - Percentage of Catheters Used Per Participant Procedure
Description: as for outcome 6
Time Frame: Patient will be followed for minimum 12 months, maximum 14 months after index Phased RFA
Population: Persistent AF patients only
Measure: Number; unit: percentage of patient procedures
Arm/Group | Phased RFA System
Number analyzed (Participants) | 279
percentage of patient procedures
  Phased RFA catheters used | 100
  MAAC catheters used | 5.4
  MASC catheters used | 4.7
  Other catheters | 11.5

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) including their relatedness to the respective procedure, were documented starting from the first documented procedure until the 12-month FU (follow-up). Analysis was performed at 30 days and 12 months after procedure.
Description: For the analysis, only adjudicated Adverse Event (AE) data and coded AE data (from free text fields) were used. In addition, TIA (transient ischaemic attack)/stroke events were taken from from the general follow-up forms to calculate procedure safety.
Arm/Group | Phased RFA System
All-Cause Mortality (participants affected / at risk) | 4/1071
Serious Adverse Events (participants affected / at risk) | 42/1071
Other Adverse Events (participants affected / at risk) | 63/1071
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phased RFA System (N=1071)
Pneumothorax (General disorders) | 1
Vascular access complication (General disorders) | 14
Other diagnosis (General disorders) | 19 — Classified as other
Stroke (General disorders) | 3
Left Atrial Fibrillation (General disorders) | 3
Acute Coronary Syndrome (General disorders) | 1
Phrenic Nerve Damage (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phased RFA System (N=1071)
Vascular Access Complication (General disorders) | 7
Other (diagnosis) (General disorders) | 51 — Other
Left Atrial Fibrillation (General disorders) | 1
Acute Coronary Syndrome (General disorders) | 1
Pulmonary Vein (PV) Stenosis (General disorders) | 1
Transient Ischaemic Attack (TIA) (General disorders) | 1
Bleeding (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details are described in the project specific Publication Plan.

DOCUMENTS (2):
  • Study Protocol (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT02433613/Prot_001.pdf
  • Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT02433613/SAP_000.pdf